CLINICAL TRIAL: NCT06205979
Title: Relationship Between Dyslipidemia and The Response of Diabetic Macular Edema to Intravitreal Injection of Anti Vascular Endothelial Growth Factor Agents
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ola Gamal Amin, resident of ophthalmology at el Helal hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-12-09MS
Record Dates: First submitted 2024-01-03; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ranibizumab Injection [Lucentis] — Three consecutive monthly intravitreal injections of Ranibizumab at a dosage of 0.5mg/0.05ml were administered in a sterile manner using a 30-G needle toward the center of the vitreous at 4mm in phakic or 3.5mm in pseudo phakic eyes from the limbus.
Drug: Aflibercept Injection [Eylea] — Three consecutive monthly intravitreal injections of Aflibercept at a dosage of 2mg/0.05ml were administered in a sterile manner using a 30-G needle toward the center of the vitreous at 4mm in phakic or 3.5mm in pseudo phakic eyes from the limbus.

SUMMARY:
Diabetic retinopathy (DR) is considered the main etiology of blindness among working-age adults, and Diabetic macular edema (DME) is the main reason for vision loss related to DR . Retinal oedema is responsible for retinal micro-structural alterations, retinal atrophy of photoreceptors and ganglion cell disorders . In addition, it might be considered consensual that the best improvements in VA could be accomplished when retinal oedema is managed. In the context of a chronic and progressive disease, DME has to be faced as a state to control as effectively and rapidly as possible . Vascular endothelial growth factor (VEGF) is a protein that promotes the growth of new blood vessels. It also makes the blood vessels more leaky. Anti- VEGF medicines stop the growth of these new blood vessels. This prevents damage to the retinal light receptors and loss of central vision. The DME treatment has been shifted from the laser photocoagulation to anti-VEGF therapy . The advantages of anti-VEGF therapy in decreasing DME and improving patient's vision have been reported in many studies . Ranibizumab, in addition to aflibercept, have been reported as the first line therapies among the other anti-VEGF . There are several data demonstrating the efficiency of ranibizumab in treatment of patients with DME . On the other hand, there are studies that revealed poor response of some patients to anti-VEGF therapies even after 3 or more injections Non-modifiable risk factors for diabetic retinopathy are gender and DM duration.

Modifiable risk factors contributing to the development of diabetic retinopathy are elevated blood sugar levels, blood pressure, and dyslipidemia which is the imbalance of lipids such as cholesterol, low-density lipoprotein cholesterol, (LDL-C), triglycerides, and high-density lipoprotein (HDL). This condition can result from diet, tobacco exposure, or genetic . Hard exudates are thought to be induced by the leakage of lipids from dysfunctional retinal capillaries . Therefore, theses were formulated that higher levels of total cholesterol, LDL-C and triglycerides could be considered biomarkers of the development of hard exudates in DM patients . Aim of the work

- Correlate between dyslipidemia and the response of patients with diabetic macular oedema to intravitreal anti-VEGF injection

ELIGIBILITY:
Inclusion Criteria:

* patients with type II DM and center involving DME with central foveal thickness more than 280 um.

Exclusion Criteria:

1. Evidence of macular ischemia
2. Evidence of macular traction
3. Previous intravitreal injections
4. Previous macular laser therapy
5. Previous pars plana vitrectomy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-06-14 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
change in the best corrected visual acuity in meters | 2 months
  measure of the ability of the eye to distinguish shapes and the details of objects at a given distance with the help of corrective lenses
change in the retina and macula measurements by Optical coherence tomography (OCT) | 2 months
  assess the state of the retina and macula by measuring :
  * Average Thickness in (μm)
change in the retina and macula measurements by Optical coherence tomography (OCT) | 2 months
  assess the state of the retina and macula by measuring :
  * Center thickness in (μm)
change in the retina and macula measurements by Optical coherence tomography (OCT) | 2 months
  assess the state of the retina and macula by measuring :
  * Total volume in (mm3)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Abramoff MD, Lavin PT, Birch M, Shah N, Folk JC. Pivotal trial of an autonomous AI-based diagnostic system for detection of diabetic retinopathy in primary care offices. NPJ Digit Med. 2018 Aug 28;1:39. doi: 10.1038/s41746-018-0040-6. eCollection 2018. PMID 31304320
- [Background] Bressler SB, Ayala AR, Bressler NM, Melia M, Qin H, Ferris FL 3rd, Flaxel CJ, Friedman SM, Glassman AR, Jampol LM, Rauser ME; Diabetic Retinopathy Clinical Research Network. Persistent Macular Thickening After Ranibizumab Treatment for Diabetic Macular Edema With Vision Impairment. JAMA Ophthalmol. 2016 Mar;134(3):278-85. doi: 10.1001/jamaophthalmol.2015.5346. PMID 26746868
- [Background] Ashraf M, Souka A, Adelman R. Predicting outcomes to anti-vascular endothelial growth factor (VEGF) therapy in diabetic macular oedema: a review of the literature. Br J Ophthalmol. 2016 Dec;100(12):1596-1604. doi: 10.1136/bjophthalmol-2016-308388. Epub 2016 May 26. PMID 27231313
- [Background] Katz G, Moisseiev E, Goldenberg D, Moisseiev J, Lomnicky Y, Abend Y, Treister G, Levkovitch-Verbin H. Ranibizumab for persistent diabetic macular edema after bevacizumab treatment. Eur J Ophthalmol. 2017 Mar 10;27(2):210-214. doi: 10.5301/ejo.5000838. Epub 2016 Jul 18. PMID 27445070